CLINICAL TRIAL: NCT03647930
Title: The Effect of Arista on Post-Operative Bleeding and Wound Drainage Following Mastectomy: A Prospective Randomized Trial
Brief Title: The Effect of Arista on Post-Operative Bleeding and Wound Drainage Following Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Health University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHUMC 2012.05.05
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Seroma
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): Application of Microporous Polysaccharide Hemospheres (MPH)
  Interventions: Device: Microporous Polysaccharide Hemospheres (MPH)
- Control (No Intervention): No MPH

INTERVENTIONS:
Device: Microporous Polysaccharide Hemospheres (MPH) — Microporous Polysaccharide Hemospheres (MPH)
  Arms: Intervention

SUMMARY:
Study aim was to evaluate topical MPH on the risk of post-mastectomy seroma formation as measured by total drain output and total drain days.

DETAILED DESCRIPTION:
Seroma formation is the most common complication after mastectomy and places patients at risk of associated morbidities. Microporous Polysaccharide Hemospheres (MPH) consists of hydrophilic, plant based, polysaccharide particles and is currently used as an absorbable hemostatic agent. An animal model evaluating MPH and seroma formation after mastectomy with axillary lymph node dissection showed a significant decrease in seroma volume. Study aim was to evaluate topical MPH on the risk of post-mastectomy seroma formation as measured by total drain output and total drain days.

Prospective randomized single-blinded clinical trial of patients undergoing mastectomy for the treatment of breast cancer. MPH was applied to the surgical site in the study group and no application in the control group.

Fifty patients were enrolled; eight were excluded due to missing data. Forty-two patients were evaluated, control (n=21) vs. MPH (n=21). No difference was identified between the two groups regarding demographics, tumor stage, total drain days, total drain output, number of clinic visits, or complication rates. On a subset analysis, body mass index (BMI) greater than 30 was identified as an independent risk factor for high drain output. Post hoc analyses of MPH controlling for BMI also revealed no statistical difference.

Unlike the data presented in an animal model, no difference was demonstrated in the duration and quantity of serosanguinous drainage related to the use of MPH in patients undergoing mastectomy for the treatment of breast cancer. BMI greater than 30 was identified as an independent risk factor for high drain output and this risk was not affected by MPH use.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Undergoing simple mastectomy with or without sentinel lymph nodes biopsy OR modified radical mastectomy for the treatment of breast cancer

Exclusion Criteria:

* Undergoing partial mastectomy
* Sentinel lymph node biopsy requiring conversion to axillary lymph node dissection
* Immediate reconstructive surgery
* Systemic anticoagulation
* Choosing not to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2015-03-06 (Actual); Study Completion 2015-03-06 (Actual)

PRIMARY OUTCOMES:
Total Drain Days | 23 Days
  Time to Drain Removal
Total Drain Output | 23 Days
  Total Drain Output in mL

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Health University Medical Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suarez-Kelly LP, Pasley WH, Clayton EJ, Povoski SP, Carson WE, Rudolph R. Effect of topical microporous polysaccharide hemospheres on the duration and amount of fluid drainage following mastectomy: a prospective randomized clinical trial. BMC Cancer. 2019 Jan 23;19(1):99. doi: 10.1186/s12885-019-5293-1. PMID 30674296